CLINICAL TRIAL: NCT02747511
Title: Intravenous Haloperidol for the Treatment of Headache in the Emergency Department
Brief Title: IV Haloperidol for the Treatment of Headache in the ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Michigan University School of Medicine (Other)
Responsible Party: Principal Investigator, Jessica McCoy, Clinical Associate Professor, Western Michigan University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMH-2015-0811
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Headache; Migraine Disorders
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Haloperidol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Haloperidol (Active Comparator)
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol
  Arms: Haloperidol
Drug: Placebo
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
Single center, double-blind, randomized, placebo-controlled trial evaluating analog pain scores in patients who present to the emergency department (ED) with a complaint of headache. A total of 150 patients age 13-55 presenting to the emergency department with headache will be enrolled from October 2015 - October 2016. Patients will be randomized and pain scores and side effects will be recorded at 0, 30, 60, and 90 minutes. Follow-up will be performed by telephone at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients that complain of headache or migraine
* Males and females age 13-55
* English is primary language

Exclusion Criteria:

* Abnormal blood pressure (>200/100)
* Sudden rapid onsent (normal to worst pain in minutes)
* Fever
* Trauma
* Any history of masses, strokes, head injury or other causes of abnormal anatomy
* QT greater than 450 ms on EKG
* Allergy to Haldon
* Any altered mental status (GCS <15)
* Pregnancy
* Any abnormalities on neurologic exam
* Any clinician concern that would require CT scan of brain
* Any prisoner or ward of state

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
>50% reduction in pain per Visual Analog Scale (VAS) | 90 minute interval

REFERENCES:
- [Derived] McCoy JJ, Aldy K, Arnall E, Petersen J. Treatment of Headache in the Emergency Department: Haloperidol in the Acute Setting (THE-HA Study): A Randomized Clinical Trial. J Emerg Med. 2020 Jul;59(1):12-20. doi: 10.1016/j.jemermed.2020.04.018. Epub 2020 May 10. PMID 32402480